CLINICAL TRIAL: NCT00191243
Title: A Randomized Phase II Study Comparing Single-Agent Docetaxel to Alternating Docetaxel-Gemcitabine as Primary Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: Docetaxel vs. Docetaxel-Gemcitabine in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5758; B9E-MC-S241 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Gemcitabine; Drug: docetaxel
- B (Experimental)
  Interventions: Drug: Gemcitabine; Drug: docetaxel

INTERVENTIONS:
Drug: Gemcitabine — A: second line therapy - 1000 mg/m2, IV, day 1 and day 8 q 21 days until disease progression
  B: 1000 mg/m2, IV, day 1 and day 8 q 21 days, until treatment failure
  Other Names: LY188011; Gemzar
Drug: docetaxel — A: 80 mg/m2, IV, q 21 days until treatment failure followed by second line single agent gemcitabine
  B: 80 mg/m2, IV, q 21 days until treatment failure

SUMMARY:
Randomized,non-blinded,multi-center study in patients with metastatic breast cancer.Patients will be treated with docetaxel or docetaxel-gemcitabine.

Aim of the study is to assess the optimal dosage and safety in this setting.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified diagnosis of breast carcinoma, at first diagnosis
* restricted previous adjuvant chemotherapy (completed >6 months prior the study)
* measurable and/or non-measurable disease
* previous radiotherapy is allowed if:terminated at least 10 days prior the sudy therapy, at least one target lesion for evaluation of tumor response has not been irradiated
* performance status 0-2 (WHO, Zubrod)
* adequate bone marrow reserve defined
* adequate liver / renal functions defined

Exclusion Criteria:

* any prior systematic chemotherapy for metastatic breast cancer
* expected survival time less than 12 weeks
* past or current history of malignant neoplasm other than breast carcinoma

  * except for cured non-melanoma skin cancer or curatively treated in situ carcinoma of the cervix uteri
* known brain metastases/leptomeningeal involvement
* active uncontrolled infection
* symptomatic peripheral neuropathy > grade 2 according to NCI
* patients whose lesions are assessable only by radionuclide scan or patients with sclerotic bone lesions as the only site of disease
* concomitant illness that is contraindication to the use of corticosteroids
* other concomitant serious illness or medical condition, which may worsen due to the treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2002-03; Primary Completion 2007-08 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTTF) | baseline to stopping treatment

SECONDARY OUTCOMES:
Response rate | baseline to measured progressive disease
Duration of response | time of response to progressive disease
Overall survival | baseline to date of death from any cause
Time to progressive disease | baseline to measured progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Finland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hämeenlinna
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jyväskylä
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lappeenranta
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pikonlinna
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pori
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Joensuu H, Sailas L, Alanko T, Sunela K, Huuhtanen R, Utriainen M, Kokko R, Bono P, Wigren T, Pyrhonen S, Turpeenniemi-Hujanen T, Asola R, Leinonen M, Hahka-Kemppinen M, Kellokumpu-Lehtinen P. Docetaxel versus docetaxel alternating with gemcitabine as treatments of advanced breast cancer: final analysis of a randomised trial. Ann Oncol. 2010 May;21(5):968-73. doi: 10.1093/annonc/mdp397. Epub 2009 Oct 9. PMID 19819914
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com